CLINICAL TRIAL: NCT02726789
Title: Therapeutic Safety and Efficacy of Combination Treatment With REP 2139-Ca and Pegasys in Patients With Chronic Hepatitis B
Brief Title: Combination Treatment With REP 2139-Ca and Pegasys in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Replicor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REP 201
Record Dates: First submitted 2016-03-18; First posted 2016-04-04 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2017-02

CONDITIONS: Hepatitis B, Chronic
Keywords: nucleic acid polymer REP 2139 HBsAg hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Patients either treatment naive or with HBV DNA controlled with entecavir receive REP 2139-Ca in combination with pegylated interferon. Only patients receiving entecavir at enrollment continue to receive entecavir during treatment in the study.
  Interventions: Drug: REP 2139-Ca; Drug: pegylated interferon; Drug: entecavir

INTERVENTIONS:
Drug: REP 2139-Ca — the nucleic acid polymer REP 2139 formulated as a calcium chelate complex
Drug: pegylated interferon — immunotherapy
  Other Names: pegylated interferon alpha 2a, Pegasys(R)
Drug: entecavir — local generic entecavir
  Other Names: local generic entecavir

SUMMARY:
The REP 201 protocol is a small exploratory study assessing the antiviral effects and tolerability of REP 2139-Ca when used with a full course of pegylated interferon (48 weeks) in treatment naive patients or in patients already receiving entecavir and continuing entecavir with treatment.

DETAILED DESCRIPTION:
Chronic hepatitis B is a long term condition caused by infection of the body with the hepatitis B virus (HBV). This infection often results in inflammation or scarring of the liver and can eventually lead to liver cirrhosis and liver failure. These infections are also one of the major causes of the development of hepatocellular carcinoma (liver cancer).

Although some drugs have been approved to treat chronic hepatitis B infections, they do not provide a complete cure except in rare cases (a cure generally means that a person loses the hepatitis B virus from the blood and the liver and develops a durable immunological control of subsequent HBV infection). However, these drugs do significantly decrease the risk of liver damage and liver cancer arising from the presence of a chronic liver infection by slowing or stopping the production of infectious virus. Thus the primary problem associated with currently available drugs is the lack of clearance of the virus from the hepatocytes which necessitates long term treatment with these drugs. There is clearly a need to identify new drugs that can benefit patients with chronic hepatitis B infections. Nucleic acid-based polymers (NAPs) are a new class of broad-spectrum antiviral compounds which act against HBV infection by blocking the release of the surface antigen protein (HBsAg) from infected hepatocytes.

Current interim data analysis from the REP 102 assessing the activity of the NAP REP 9AC' (REP 2139, given as a calcium chelate complex [REP 2139-Ca]) in patients with chronic HBV infection indicates the following:

1. REP 2139-Ca is generally well tolerated and patients tolerate short term combined treatment (13-26 weeks) of pegylated interferon and / or thymosin alpha
2. REP 2139-Ca has achieved serum HBsAg reduction or clearance 9 of 9 patients receiving combined therapy.
3. Appearance of substantial titers of serum anti-HBs occur with the addition of immunotherapy.
4. After all treatment is withdrawn, 8 / 9 patients achieved HBV DNA < 116 copies / ml (LLOQ of the Roche Cobas platform) and sustained suppression of viremia (HBV DNA < 1000 cpm, HBsAg < 1 IU / ml) for a period of greater than 1 year was observed in four patients.

This exploratory study is designed to examine if REP 2139-Ca can be safely combined with a full course of pegylated interferon in treatment naive patients and in patients with previous and continuing therapy with entecavir and that similar antiviral effects can be observed as in the previous REP 101 and 102 protocols.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55
* HBsAg+
* Anti-HBs negative
* Patients currently receiving nucleoside based HBV polymerase inhibitors may be included in the study at the discretion of the Principle Investigator.
* HIV / hepatitis C / hepatitis delta virus negative
* Fibrosis with compensation (as determined by Fibroscan and liver enzymes)
* Non cirrhotic
* No known active cytomegalovirus infection
* Willingness to utilize adequate contraception while being treated with REP 9AC' and for 6 months following the end of treatment
* Adequate venous access allowing weekly intravenous therapies and blood tests

Exclusion Criteria:

* Evidence of cardiovascular disease
* Autoimmune hepatitis
* Presence of Wilson's disease
* Presence of severe NAFLD
* Evidence of any other co-existent liver disease
* Anti-nuclear antibody positive
* Ultrasonograph of hepato-biliary system: positive for cirrhosis of liver
* A history of ascites, hepatic encephalopathy or variceal hemorrhage
* Body weight > 100 kg
* Platelet count < 75,000, polymorphonuclear cell count < 1,500 or hematocrit < 33%
* alpha feto protein > 100 ng/ml or the presence of a hepatic mass suggestive of hepatocellular carcinoma .
* Bilirubin > 2.5 mg/dl
* Creatinine > 1.5 mg/dl
* Platelet count < 75,000 / cmm
* Serum albumin < 35 mg/ml
* Poorly controlled diabetes mellitus
* Another serious medical disorder
* A serious psychiatric disorder
* Uncontrolled hypertension
* A history of alcohol abuse within the last year
* The use of illicit drugs within the past two years
* Inability to provide informed consent
* Positive pregnancy test
* Breastfeeding
* Inability or unwillingness to provide weekly blood samples
* Poor venous access making IV infusion too difficult

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mamun Al-Mahtab, MD, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers inhibit duck hepatitis B virus infection in vitro. Antimicrob Agents Chemother. 2013 Nov;57(11):5291-8. doi: 10.1128/AAC.01003-13. Epub 2013 Aug 12. PMID 23939902
- [Background] Noordeen F, Vaillant A, Jilbert AR. Nucleic acid polymers prevent the establishment of duck hepatitis B virus infection in vivo. Antimicrob Agents Chemother. 2013 Nov;57(11):5299-306. doi: 10.1128/AAC.01005-13. Epub 2013 Aug 12. PMID 23939904
- [Background] Noordeen F, Scougall CA, Grosse A, Qiao Q, Ajilian BB, Reaiche-Miller G, Finnie J, Werner M, Broering R, Schlaak JF, Vaillant A, Jilbert AR. Therapeutic Antiviral Effect of the Nucleic Acid Polymer REP 2055 against Persistent Duck Hepatitis B Virus Infection. PLoS One. 2015 Nov 11;10(11):e0140909. doi: 10.1371/journal.pone.0140909. eCollection 2015. PMID 26560490

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Patients to receive REP 2139-Ca in combination with pegylated interferon. Participants included in this study are either entecavir naive OR have prior exposure to entecavir.
Period: Overall Study
Arm/Group | Experimental
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Participants receive REP 2139-Ca in combination with pegylated interferon. Participants included in this study are either entecavir naive OR have prior exposure to entecavir.
  REP 2139-Ca: the nucleic acid polymer REP 2139 formulated as a calcium chelate complex
  pegylated interferon: immunotherapy
  Participants receiving entecavir at the start of therapy continue to receive entecavir during experimental therapy.
Arm/Group | Experimental
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (3.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  Bangladesh | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Treatment Emergent Laboratory Test Abnormalities or Adverse Events.
Description: To record side effects, symptoms and adverse effects of exposure to REP 2139-Ca when combined pegylated interferon.
Time Frame: 48 weeks (treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Participants receive REP 2139-Ca in combination with pegylated interferon. Participants included in this study are either entecavir naive OR have prior exposure to entecavir.
  REP 2139-Ca: the nucleic acid polymer REP 2139 formulated as a calcium chelate complex
  pegylated interferon: immunotherapy
  Participants receiving entecavir at the start of experimental therapy continue to receive entecavir throughout experimental therapy.
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Number of Patients Experiencing Reductions in Serum HBsAg
Description: To assess antiviral activity of REP 2139-Ca when combined with pegylated interferon on serum HBsAg.
Time Frame: 48 weeks (treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Participants receive REP 2139-Ca in combination with pegylated interferon. Participants included in this study are either entecavir naive OR have prior exposure to entecavir.
  REP 2139-Ca: the nucleic acid polymer REP 2139 formulated as a calcium chelate complex
  pegylated interferon: immunotherapy
  Partiipants receiving entecavir at the start of experimental therapy continue to receive entecavir throughout experimental therapy.
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 5

3. Secondary Outcome: Number of Patients Experiencing Reductions in Serum HBV DNA
Description: To assess antiviral activity of REP 2139-Ca when combined with pegylated interferon on serum HBV DNA.
Time Frame: 48 weeks (treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 5

4. Secondary Outcome: Number of Patients Experiencing Serum Anti-HBs > 10 mIU / ml
Description: To assess antiviral activity of REP 2139-Ca when combined with pegylated interferon on anti-HBsAg antibody titer.
Time Frame: 48 weeks (treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 3 years
Description: Weekly patient surveillance during therapy, every 1-8 weeks during follow-up
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=5)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) — Nephrotic syndrome occurred at week 38 exposure secondary to facial edema presence of urine albumin . Pegasys® therapy was halted early in this patient who recovered during the follow-up with supportive therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=5)
ALT elevation (Hepatobiliary disorders) | 5 (5) — Transient, self resolving elevations in serum ALT not accompanied by elevation in bilirubin or INR.
Weakness (General disorders) | 5 (23)
Reduced appetite (General disorders) | 5 (21)
Hairloss (General disorders) | 5 (13)
Nausea (Gastrointestinal disorders) | 5 (8)
Asthenia (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Abdominal cramping (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Dusgeusia (Gastrointestinal disorders) | 5 (9)
Chest pain (Cardiac disorders) | 2 (2)
Pain / tingling in periphery (Nervous system disorders) | 5 (11)
Fever (General disorders) | 3 (6)
Generalized body ache (General disorders) | 2 (5)
Weight loss (General disorders) | 5 (8)
AST elevation (Hepatobiliary disorders) | 5 (5) — Transient, self resolving elevations in serum AST not accompanied by elevation in bilirubin or INR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No